CLINICAL TRIAL: NCT01326962
Title: Tocilizumab Efficacy and Safety in RA Patients After Inadequate Response to DMARDs or Anti-TNF
Brief Title: A Study of RoActemra/Actemra (Tocilizumab) in Patients With Rheumatoid Arthritis Who Have an Inadequate Response to DMARDs or Anti-TNF
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML22726
Record Dates: First submitted 2011-03-07; First posted 2011-03-31 (Estimated); Results first posted 2016-03-28 (Estimated); Last update posted 2017-08-16 (Actual); Status verified 2017-07

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — tocilizumab

ARMS (1):
- Single Arm (Experimental)
  Interventions: Drug: tocilizumab [RoActemra/Actemra]

INTERVENTIONS:
Drug: tocilizumab [RoActemra/Actemra] — 8 mg/kg (max. 800 mg) iv every 4 weeks, 6 infusions

SUMMARY:
This open-label, single arm study will evaluate the safety and efficacy of RoActemra/Actemra (tocilizumab) in patients with active, moderate to severe rheumatoid arthritis who have an inadequate response to disease-modifying antirheumatic drugs (DMARDs) or anti-TNF. Patients will receive RoActemra/Actemra at a dose of 8 mg/kg (max 800 mg) intravenously every 4 weeks for a total of 6 infusions. Non-biologic DMARD therapy may be continued throughout the study. Anticipated time on study treatment is 24 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, >/= 18 years of age
* Active moderate to severe rheumatoid arthritis of >/= 6 months duration
* >/=1 non-biologic DMARD and/or anti-TNF therapy at stable dose for >/=8 weeks at any time prior to study treatment
* Inadequate clinical response to non-biologic DMARD or anti-TNF therapy
* Oral corticosteroids must be at stable dose for at least 25 out of 28 days prior to first dose of study drug

Exclusion Criteria:

* Pregnant or lactating women
* Major surgery (including joint surgery) within 8 weeks prior to screening or major surgery planned within 6 months of enrolment
* Rheumatic autoimmune disease other than RA
* Functional class IV (ACR classification)
* Prior history of or current joint disease other than RA
* Intraarticular or parenteral corticosteroids within 6 weeks prior to baseline
* Previous treatment with RoActemra/Actemra
* Known active current or history of recurrent infection
* History of or currently active primary or secondary immunodeficiency
* Active tuberculosis requiring treatment within the previous 3 years
* Positive for HIV

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2011-11-30 (Actual); Primary Completion 2013-05-12 (Actual); Study Completion 2013-05-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (4):
- Saudi Arabia (4):
  - King Fahad Specialist Hospital; Oncology, Dammam
  - King Abdulaziz University Hospital, Jeddah
  - Heraa General Hospital; Rheumatology, Mecca
  - King Fahad Medical City; Gastroentrology, Riyadh

REFERENCES:
- [Derived] Abdulkader OAF, Qushmaq K, Aljishi F. Tocilizumab efficacy and safety in rheumatoid arthritis patients after inadequate response to disease-modifying anti-rheumatic drugs oranti-tumor necrosis factor. Ann Saudi Med. 2016 May-Jun;36(3):190-6. doi: 10.5144/0256-4947.2016.190. PMID 27236390

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 3 centers ( 1 center was prematurely terminated) across the Kingdom of Saudi Arabia from 02 November 2011 to 12 May 2013.
Groups:
- Tocilizumab: Participants received Tocilizumab 8 milligram per kilogram (mg/kg) intravenously (IV) every 4 weeks for a total of 6 infusions up to Week 20. A follow-up visit at Week 24 was planned, after which evaluation of responders was done. Good/moderate EULAR responders continued receiving Tocilizumab every 4 weeks, till 1 year treatment or commercial availability.
Period: Overall Study
Arm/Group | Tocilizumab
Started | 28
Completed | 21
Not Completed | 7
Not completed — Adverse Event | 1
Not completed — Withdrawal by Subject | 1
Not completed — Lost to Follow-up | 3
Not completed — Other | 2

BASELINE CHARACTERISTICS:
Arm/Group | Tocilizumab
Number analyzed (Participants) | 28
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.1 (12.40)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26
  Male | 2

OUTCOME MEASURES:

1. Primary Outcome: Disease Activity as Measured by Disease Activity Score 28 (DAS28)
Description: The DAS28 is a combined index for measuring disease activity in rheumatoid arthritis (RA). The index includes swollen (range 0-28) and tender (range 0-28) joint counts, acute phase response (erythrocyte sedimentation rate [ESR] in millimeters per hour [mm/hr]), and general health status (participant global assessment of disease activity using visual analog scale [VAS], range 1-100 mm). DAS28, which uses a 28-joint count, is derived from the original DAS, which includes a 44-swollen joint count. The DAS28 scale ranges from 0 to 10, where higher scores represent higher disease activity.
Time Frame: Up to 1 year
Population: The intent-to-treat population (ITT) consisted of all consented participants enrolled in the study, who had received any part of an infusion of study medication. Where, 'n' is equal to (=) number of participants analyzed at particular point of time.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Groups:
- Tocilizumab: Participants received Tocilizumab 8 mg/kg IV every 4 weeks for a total of 6 infusions up to Week 20.
Arm/Group | Tocilizumab
Number analyzed (Participants) | 28
units on a scale
  Baseline (n=28) | 5.4 [4.1 to 7.9]
  Visit 3 (n=27) | 3.5 [1.9 to 5.7]
  Visit 4 (n= 26) | 2.8 [0.9 to 5.5]
  Visit 5 (n= 25) | 2.2 [1.3 to 4.2]
  Visit 6 (n= 25) | 1.9 [0.4 to 4.6]
  Visit 7 (n= 25) | 1.7 [0.5 to 2.8]
  Visit 8 (n= 23) | 1.7 [0.5 to 3.4]
  Visit 9 (n= 21) | 1.9 [0.0 to 3.7]
  Visit 10 (n= 22) | 1.7 [0.0 to 3.2]
  Visit 11 (n= 21) | 2.0 [0.1 to 5.0]
  Visit 12 (n= 17) | 2.3 [1.0 to 4.4]
  Visit 13 (n= 13) | 2.1 [0.1 to 3.6]
  Visit 14 (n= 6) | 1.5 [0.1 to 5.6]

2. Primary Outcome: Number of Participants Who Achieved Remission (DAS28 < 2.6)
Description: The DAS28 is a combined index for measuring disease activity in RA. The index includes swollen (range 0-28) and tender (range 0-28) joint counts, acute phase response (ESR in mm/hr), and general health status (participant global assessment of disease activity using VAS, range 1-100 mm). DAS28, which uses a 28-joint count, is derived from the original DAS, which includes a 44-swollen joint count. The DAS28 scale ranges from 0 to 10, where higher scores represent higher disease activity.
Time Frame: Up to 1 year
Population: ITT consisted of all consented participants enrolled in the study, who had received any part of an infusion of study medication. Where, 'n' = number of participants analyzed at particular point of time.
Measure: Number; unit: participants
Arm/Group | Tocilizumab
Number analyzed (Participants) | 27
participants
  Visit 3 (n=27) | 3
  Visit 4 (n=26) | 7
  Visit 5 (n=25) | 12
  Visit 6 (n=25) | 14
  Visit 7 (n=25) | 17
  Visit 8 (n=23) | 16
  Visit 9 (n=21) | 15
  Visit 10 (n=22) | 18
  Visit 11 (n=21) | 13
  Visit 12 (n=17) | 7
  Visit 13 (n=13) | 8
  Visit 14 (n=6) | 4

3. Primary Outcome: Time to Das28 Remission
Description: Time to DAS28 Remission was the Time in days from the first infusion of study drug to the achievement of a DAS28 score < 2.6 units. The DAS28 is a combined index for measuring disease activity in RA. The index includes swollen (range 0-28) and tender (range 0-28) joint counts, acute phase response (ESR in mm/hr), and general health status (participant global assessment of disease activity using VAS, range 1-100 mm). DAS28, which uses a 28-joint count, is derived from the original DAS, which includes a 44-swollen joint count. The DAS28 scale ranges from 0 to 10, where higher scores represent higher disease activity.
Time Frame: Up to 1 year
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Day
Arm/Group | Tocilizumab
Number analyzed (Participants) | 28
Day | 189.01 (7.053)

4. Primary Outcome: Number of Participants Who Achieved a Clinically Meaningful Improvement in DAS28 (Reduction of At Least 1.2 Units)
Description: DAS28 Clinically Significant Improvement was defined as a DAS28 score reduction of at least 1.2 units from Baseline. The DAS28 is a combined index for measuring disease activity in RA. The index includes swollen (range 0-28) and tender (range 0-28) joint counts, acute phase response (ESR in mm/hr), and general health status (participant global assessment of disease activity using VAS, range 1-100 mm). DAS28, which uses a 28-joint count, is derived from the original DAS, which includes a 44-swollen joint count. The DAS28 scale ranges from 0 to 10, where higher scores represent higher disease activity.
Time Frame: Up to 1 year
Population: ITT population consisted of all consented participants enrolled in the study, who had received any part of an infusion of study medication. Where, 'n' = number of participants analyzed at particular point of time.
Measure: Number; unit: participants
Arm/Group | Tocilizumab
Number analyzed (Participants) | 28
participants
  Visit 3 (n=27) | 21
  Visit 4 (n=26) | 20
  Visit 5 (n=25) | 20
  Visit 6 (n=25) | 22
  Visit 7 (n=25) | 21
  Visit 8 (n=23) | 20
  Visit 9 (n=21) | 19
  Visit 10 (n=22) | 20
  Visit 11 (n=21) | 17
  Visit 12 (n=17) | 12
  Visit 13 (n=13) | 11
  Visit 14 (n=6) | 4

5. Primary Outcome: Number of Participants Who Achieved Low Disease Activity (DAS28 < 3.2)
Description: DAS28 low disease activity was defined as a DAS28 score reduction of at least 3.2 units from Baseline. The DAS28 is a combined index for measuring disease activity in RA. The index includes swollen (range 0-28) and tender (range 0-28) joint counts, acute phase response (ESR in mm/hr), and general health status (participant global assessment of disease activity using VAS, range 1-100 mm). DAS28, which uses a 28-joint count, is derived from the original DAS, which includes a 44-swollen joint count. The DAS28 scale ranges from 0 to 10, where higher scores represent higher disease activity.
Time Frame: Up to 1 year
Population: as for outcome 4
Measure: Number; unit: participants
Arm/Group | Tocilizumab
Number analyzed (Participants) | 27
participants
  Visit 3 (n=27) | 7
  Visit 4 (n=26) | 9
  Visit 5 (n= 25) | 7
  Visit 6 (n=25) | 7
  Visit 7 (n=25) | 4
  Visit 8 (n= 23) | 3
  Visit 9 (n=21) | 3
  Visit 10 (n=22) | 2
  Visit 11 (n=21) | 2
  Visit 12 (n=17) | 4
  Visit 13 (n=13) | 1
  Visit 14 (n=6) | 0

6. Primary Outcome: Number of Participants Who Achieved Clinically Meaningful Health Assessment Questionnaire Response
Description: Health Assessment Questionnaire (HAQ) is a self-completed participant questionnaire specific for Rheumatoid Arthritis. It consists of 20 questions referring to 8 domains: dressing/grooming, arising, eating, walking, hygiene, reach, grip; common daily activities. Each domain has at least 2 component questions. There are 4 possible responses for each component 0=without any difficulty, 1=with some difficulty, 2=with much difficulty, and 3=unable to do. To calculate HAQ, the participant must have a domain score for at least 6 out of 8 domains. The HAQ is the sum of the scores, divided by the number of domains that have a score (in range 6-8) for a total possible score minimum/maximum 0 (best) to 3 (worst). A negative change from baseline indicated improvement. Clinically meaningful HAQ response was defined as an improvement of at least 0.22 units from baseline in the HAQ Disability Index.
Time Frame: Up to 1 year
Population: as for outcome 4
Measure: Number; unit: participants
Arm/Group | Tocilizumab
Number analyzed (Participants) | 28
participants
  Visit 3 (n=27) | 7
  Visit 4 (n=25) | 6
  Visit 5 (n= 25) | 6
  Visit 6 (n=25) | 7
  Visit 7 (n=25) | 6
  Visit 8 (n= 23) | 4
  Visit 9 (n=21) | 5
  Visit 10 (n=22) | 4
  Visit 11 (n=21) | 2
  Visit 12 (n=17) | 4
  Visit 13 (n=12) | 3

7. Primary Outcome: Changes in Participant's Fatigue Assessed Using the Mean FACIT-Fatigue Score
Description: The FACIT-Fatigue score was calculated according to a 13-item questionnaire that assesses self-reported fatigue and its impact upon daily activities and function. Participants scored each item on a 5-point scale: 0 (Not at all) to 4 (Very much). The larger the participant's response to the questions (with the exception of 2 negatively stated), the greater the participants fatigue. For all questions, except for the 2 negatively stated ones, the code was reversed and a new score was calculated as (4 minus the participant's response). The sum of all responses resulted in the FACIT-Fatigue score for a total possible score of 0 (worse score) to 52 (better score).
Time Frame: Up to 1 year
Population: as for outcome 4
Measure: Number; unit: Units on a scale
Arm/Group | Tocilizumab
Number analyzed (Participants) | 28
Units on a scale
  Visit 3 (n=27) | 23.5
  Visit 4 (n=26) | 24.1
  Visit 5 (n= 25) | 23.6
  Visit 6 (n=25) | 24.0
  Visit 7 (n=25) | 21.6
  Visit 8 (n= 23) | 22.0
  Visit 9 (n=21) | 19.1
  Visit 10 (n=22) | 22.3
  Visit 11 (n=21) | 27.8
  Visit 12 (n=17) | 27.3
  Visit 13 (n=13) | 26.6
  Visit 14 (n=6) | 25.6

8. Primary Outcome: Change in Fatigue as Measured Using the Fatigue Visual Analog Scale
Description: The VAS for Fatigue (VAS-F) consists of a 100 mm line, with 0 (No Fatigue) on one end, and 100 (Extreme Fatigue) on the other end, which a participant marks to indicate how much fatigue he or she feels. The marked point in mm is converted into a numeric value from 0 to 100, where 0=no fatigue and 100=maximum fatigue. Increasing numbers=increasing fatigue.
Time Frame: Up to 1 year
Population: as for outcome 4
Measure: Number; unit: units on a scale
Arm/Group | Tocilizumab
Number analyzed (Participants) | 28
units on a scale
  Visit 3 (n=27) | 38.1
  Visit 4 (n=26) | 32.3
  Visit 5 (n= 25) | 29.0
  Visit 6 (n=25) | 20.1
  Visit 7 (n=25) | 14.4
  Visit 8 (n= 23) | 18.0
  Visit 9 (n=21) | 13.1
  Visit 10 (n=22) | 20.7
  Visit 11 (n=21) | 19.1
  Visit 12 (n=17) | 23.9
  Visit 13 (n=13) | 26.3
  Visit 14 (n=6) | 32.0

9. Secondary Outcome: Number of Participants With Any Adverse Event and Serious Adverse Event
Description: An adverse event (AE) is defined as any unfavourable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. A serious adverse event (SAE) is defined as any untoward medical occurrence that, at any dose, results in death, is life threatening, requires hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect, or is a significant medical event.
Time Frame: Up to 1 year
Population: Safety population included all participants who had received at least one dose of study medication.
Measure: Number; unit: participants
Arm/Group | Tocilizumab
Number analyzed (Participants) | 28
participants
  Any AE | 4
  Any SAE | 2

10. Secondary Outcome: Number of Participants With AE or SAE Related Discontinuation of Tocilizumab
Description: It included participants who discontinued from the study due to occurrence of AE or SAE.
Time Frame: Up to 1 year
Population: Safety population included all participants who had received at least one dose of study medication.
Measure: Number; unit: participants
Arm/Group | Tocilizumab
Number analyzed (Participants) | 28
participants | 2

11. Secondary Outcome: Number of Participants Who Achieved ACR20, ACR50, ACR70 and ACR90 Response
Description: ACR20, ACR50, ACR70, and ACR90 are defined as greater than or equal to (≥)20 percent (%), ≥50%, ≥70%, or ≥90% improvement, respectively, in swollen joint count (SJC; 66 joints) and tender joint count (TJC; 68 joints). It also comprises ≥20%, ≥50%, ≥70%, or ≥90% improvement, respectively, in 3 of the following 5 assessments: Patient's Global Assessment of Pain (VAS); Patient's Global Assessment of Disease Activity (VAS); Investigator/Physician's Global Assessment of Disease Activity (VAS); participant's assessment of disability measured by the Health Assessment Questionnaire Disability Index (HAQ-DI); or acute phase reactant (ESR or C-reactive protein [CRP]).
Time Frame: Up to 1 year
Population: as for outcome 4
Measure: Number; unit: participants
Arm/Group | Tocilizumab
Number analyzed (Participants) | 28
participants
  ACR20: Visit 3 (n=27) | 3
  ACR20: Visit 4 (n=26) | 4
  ACR20:Visit 5 (n=25) | 1
  ACR20: Visit 6 (n=25) | 1
  ACR20: Visit 7 (n=25) | 0
  ACR20: Visit 8 (n=23) | 0
  ACR20: Visit 9 (n=21) | 0
  ACR20: Visit 10 (n=22) | 0
  ACR20: Visit 11 (n=21) | 2
  ACR20: Visit 12 (n=17) | 1
  ACR20: Visit 13 (n=13) | 0
  ACR20: Visit 14 (n=6) | 0
  ACR50: Visit 3 (n=27) | 11
  ACR50: Visit 4 (n=26) | 7
  ACR50:Visit 5 (n=25) | 1
  ACR50: Visit 6 (n=25) | 1
  ACR50: Visit 7 (n=25) | 2
  ACR50: Visit 8 (n=23) | 1
  ACR50: Visit 9 (n=21) | 1
  ACR50: Visit 10 (n=22) | 1
  ACR50: Visit 11 (n=21) | 0
  ACR50: Visit 12 (n=17) | 0
  ACR50: Visit 13 (n=13) | 1
  ACR50: Visit 14 (n=6) | 1
  ACR70: Visit 3 (n=27) | 7
  ACR70: Visit 4 (n=26) | 10
  ACR70:Visit 5 (n=25) | 14
  ACR70: Visit 6 (n=25) | 8
  ACR70: Visit 7 (n=25) | 3
  ACR70: Visit 8 (n=23) | 6
  ACR70: Visit 9 (n=21) | 5
  ACR70: Visit 10 (n=22) | 6
  ACR70: Visit 11 (n=21) | 6
  ACR70: Visit 12 (n=17) | 5
  ACR70: Visit 13 (n=13) | 5
  ACR70: Visit 14 (n=6) | 0
  ACR90: Visit 3 (n=27) | 2
  ACR90: Visit 4 (n=26) | 3
  ACR90:Visit 5 (n=25) | 8
  ACR90: Visit 6 (n=25) | 13
  ACR90: Visit 7 (n=25) | 18
  ACR90: Visit 8 (n=23) | 15
  ACR90: Visit 9 (n=21) | 14
  ACR90: Visit 10 (n=22) | 14
  ACR90: Visit 11 (n=21) | 12
  ACR90: Visit 12 (n=17) | 10
  ACR90: Visit 13 (n=13) | 5
  ACR90: Visit 14 (n=6) | 3

12. Secondary Outcome: Number of Participants With C-Reactive Protein Abnormality
Description: CRP is a biological marker of inflammation. A reduction in CRP indicates improvement. It is measured in milligram per liter (mg/L).
Time Frame: Up to 1 year
Population: as for outcome 4
Measure: Number; unit: mg/L
Arm/Group | Tocilizumab
Number analyzed (Participants) | 28
mg/L
  Baseline (n=28) | 16
  Visit 3 (n=27) | 8
  Visit 4 (n=26) | 7
  Visit 5 (n=25) | 2
  Visit 6 (n=25) | 5
  Visit 7 (n=25) | 6
  Visit 8 (n=23) | 7
  Visit 9 (n=21) | 7
  Visit 10 (n=22) | 9
  Visit 11 (n=21) | 9
  Visit 12 (n=17) | 8
  Visit 13 (n=13) | 7
  Visit 14 (n=6) | 2

13. Secondary Outcome: Number of Participants With Erythrocyte Sedimentation Rate Abnormality
Description: ESR is an acute phase reactant and is a measure of inflammation. It is measured in millimeter per hour (mm/hr).
Time Frame: Up to 1 year
Population: as for outcome 4
Measure: Number; unit: participants
Arm/Group | Tocilizumab
Number analyzed (Participants) | 28
participants
  Baseline (n=28) | 13
  Visit 3 (n=27) | 5
  Visit 4 (n=26) | 3
  Visit 5 (n=25) | 1
  Visit 6 (n=25) | 0
  Visit 7 (n=25) | 1
  Visit 8 (n=23) | 2
  Visit 9 (n=21) | 3
  Visit 10 (n=22) | 0
  Visit 11 (n=21) | 0
  Visit 12 (n=17) | 0
  Visit 13 (n=13) | 2
  Visit 14 (n=6) | 1

ADVERSE EVENTS:
Time Frame: Up to 1 Year
Description: All participants enrolled were included in the safety analysis.
Arm/Group | Tocilizumab
Serious Adverse Events (participants affected / at risk) | 2/28
Other Adverse Events (participants affected / at risk) | 4/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tocilizumab (N=28)
Hypotension (Vascular disorders) | 1
Skin Rash (Skin and subcutaneous tissue disorders) | 1
Neutropenia (Blood and lymphatic system disorders) | 1
Thrombocytpenia (Blood and lymphatic system disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Tocilizumab (N=28)
Hypertension (Vascular disorders) | 1
Neutropenia (Blood and lymphatic system disorders) | 1
Low hemoglobin (Blood and lymphatic system disorders) | 1
Low red blood cells (Blood and lymphatic system disorders) | 1
Epistaxis (Blood and lymphatic system disorders) | 1
Urinary tract infection (Infections and infestations) | 1
Diplopia (Eye disorders) | 1
Dry eye (Eye disorders) | 1
Infusion site pain (General disorders) | 1
Headache & dizziness (General disorders) | 1
Headache & generalized body ache (General disorders) | 1
Fibromyalgia (Musculoskeletal and connective tissue disorders) | 1
Low back pain (Musculoskeletal and connective tissue disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Flu (Respiratory, thoracic and mediastinal disorders) | 1
Hyponatremia (Metabolism and nutrition disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.